CLINICAL TRIAL: NCT00878293
Title: A Randomized Phase IIa Trial Evaluating the Safety and Efficacy of a New Centrally Acting Analgesic in Subjects With Pain Due to Diabetic Polyneuropathy
Brief Title: Painful Diabetic Polyneuropathy Trial With a New Centrally Acting Analgesic
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tris Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 449723
Record Dates: First submitted 2009-04-03; First posted 2009-04-08 (Estimated); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Diabetic Polyneuropathy
Keywords: analgesic; diabetes mellitus; chronic neuropathic pain; painful polyneuropathy caused by diabetes mellitus type I or II
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- A (Experimental): Dose 1, 40 µg
  Interventions: Drug: GRT6005
- B (Experimental): Dose 2, 120 µg
  Interventions: Drug: GRT6005
- C (Experimental): Dose 3
  Interventions: Drug: GRT6005
- D (Experimental): Dose 4
  Interventions: Drug: GRT6005
- E (Experimental): Dose 5
  Interventions: Drug: GRT6005
- F (Experimental): Dose 6
  Interventions: Drug: GRT6005
- G (Experimental): Dose 7
  Interventions: Drug: GRT6005
- H (Active Comparator): Morphin
  Interventions: Drug: MS Continus®
- I (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GRT6005 — liquid formulation for oral application, 0,8 to 400 µg, single dose per day, five days
  Arms: A; B; C; D; E; F; G
Drug: MS Continus® — 60 mg, capsule, once daily
  Arms: H
Drug: Placebo — liquid formulation and capsule, once daily
  Arms: I

SUMMARY:
The purpose of this trial is to determine whether the new centrally active analgesic and MS Continus® are effective in the treatment of painful diabetic polyneuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with pain at least NRS >4 due to painful diabetic polyneuropaty.

Exclusion Criteria:

* Contraindications to, or history of allergy or hypersensitivity to morphine, fentanyl, hydrocodone, acetaminophen, heparin, polyethylene glycol 400 USP-NF or any compound planned to be used during the anesthesia, or their excipients.
* non Caucasian or Hispanic.
* Concomitant painful disease.
* Life-long history of seizure disorder or epilepsy.
* Subjects with clinical relevant cardiac and vascular diseases.
* Subjects with impaired renal function
* Subjects with impaired hepatic function
* Female subjects who are pregnant or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Average daily pain intensity | 5 days

SECONDARY OUTCOMES:
Quality of life Neuropathic pain scale Amount and first time of Rescue medication Adverse events, ECG, Laboratory values | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Forst, Prof. Dr. med, Principal Investigator — IKFE, Parcusstr. 8, 55116 Mainz
Locations (4):
- Germany (3):
  - Investigator 3, Bad Oeynhausen
  - Investigator 1, Mainz
  - Investigator 2, Münster
- Investigator 4, Manchester, United Kingdom